CLINICAL TRIAL: NCT02870465
Title: K-wire Infections in Operating Room Sterility Versus Ambulatory Setting Field Sterility: A Prospective Cohort Study
Brief Title: Hand K-wire Infections in Operating Room Versus Ambulatory Setting
Status: Completed | Type: Observational
Sponsor: Horizon Health Network (Other)
Responsible Party: Principal Investigator, Don Lalonde MD, Principal Investigator, Horizon Health Network
Other Study IDs: HHN-1
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Hand Fracture; Infection Due to Internal Fixation Pin
Keywords: outpatient versus operating room; k wire infection; closed reduction internal fixation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CRIF in operating room: Patients who present with a hand fracture amendable to closed reduction internal fixation (CRIF) who are managed in the operating room.
  Interventions: Procedure: Closed Reduction Internal Fixation
- CRIF outside of operating room: Patients who present with a hand fracture amendable to closed reduction internal fixation (CRIF) who are managed outside of the operating room (i.e.: in clinical setting, the emergency department or minor procedures area).
  Interventions: Procedure: Closed Reduction Internal Fixation

INTERVENTIONS:
Procedure: Closed Reduction Internal Fixation — K-wires placed percutaneously through the skin to achieve fixation of a hand after reduction of the fracture in a closed manner.

SUMMARY:
The main objective of this non-interventional, observational study is to analyze the rate and type of infection complications while performing closed reduction internal fixation (CRIF) of hand fractures in the operating room versus an ambulatory setting. The investigators will do so by prospectively collecting data on the type of fracture, handedness, co-morbidities, duration of treatment, number and type of K-wires, duration of fixation and complication rate. Patients presenting with hand fractures to the emergency room will be recruited. Patients will be recruited in multiple centres across Canada and managed according to the institutional standard. The complication type and rate will be recorded and analyzed to determine a difference of performing the procedure in the operating room or clinical setting.

DETAILED DESCRIPTION:
The main objective of this study is to analyze the rate and type of infectious complications while performing closed reduction internal fixation (CRIF) of hand fractures in the operating room versus an ambulatory setting. The investigators will do so by prospectively collecting data into a hand fracture database, recording the type of fracture, handedness, co-morbidities, duration of treatment, number of K-wires, duration of fixation and complication rate. These will be recorded on a data collection form, which will be transcribed into a password protected excel spread sheet by Dr. Lalonde. The data will be de-identified and the patients will be assigned a number to place on the data collection sheet depending on order of presentation. The investigators will include all adult patients presenting with a metacarpal or phalangeal that is amenable to CRIF with K-wires.

The investigators will recruit patients prospectively from the emergency room or clinic referrals. All patients who meet the inclusion and exclusion criteria will be asked to participate by the attending surgeon or resident. The patients will be assigned a number according to chronological presentation. The patients will be recruited from academic centers in Canada. Three centers, Halifax, Toronto and McMaster, do not perform CRIF with K-wires in a clinical setting and thus will represent the main operating room cohort. The clinical setting CRIF cohort will be comprised of patients from St. John, Calgary, Ottawa, Vancouver and St John's where CRIF of hand fractures are routinely performed under local anaesthetic and field sterility. The characteristics of the injury, fracture, timing of injury, patient comorbidities which predispose to infections, handedness, smoking status, sex and age will be recorded.

All procedures in the operating room or the clinic area will be performed under the anaesthetic that is standard in that center. A procedure will be deemed "field sterility" if the usual surgical preparation of povidone-iodine or isopropyl alcohol-chlorohexidine gluconate and sterile drape is performed with sterile gloves and masks but without surgical gowns. In the outpatient clinic area, a basic tray will be used along with the K-wire driver and wire-cutters. A mini C-arm fluoroscopy machine is used to visualize the reduction and placement of the K-wires. The patients will then be dressed with a non-antibiotic containing dressing and splinted. The surgical information such as number and type of K-wires, OR time, type of anaesthesia, place of operation, and antibiotic use will be recorded. There will be no additional pin site care offered, as there is no standard accepted method to decrease pin-tract infection. They will be followed up as per the local protocol.

The patients will be instructed that if they are concerned regarding a complication or infection that they must present to their attending surgeon or other plastic surgery colleague covering outpatient calls. They will be provided a contact number for after hours. The necessity to contact the attending team will be stressed to improve documentation of complications and ensure that the proper diagnosis of an infection will be made and appropriate antibiotic coverage started. If the patient is to present to the emergency department or family physician, improper antibiotic coverage may be started for a patient presenting with normal wound healing, which will falsely elevate the incidence of recorded hand infections. The patient will be followed until K-wire removal around 3 to 4 weeks, as per local protocol, and the duration of K-wire fixation will be recorded along with any complications.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients presenting with an acute metacarpal or phalangeal fracture amenable to closed reduction and percutaneous pinning.

Exclusion Criteria:

1. Fractures that cannot be reduced in a closed manner necessitating open reduction internal fixation
2. Multiple fractures or significant injury requiring ORIF by other means - such as plate fixation
3. Existing infection
4. Pathologic fracture
5. CRIF performed during replantation or revascularization of digit
6. Concomitant injury (tendon injury, nerve injury, soft tissue loss requiring reconstructive procedure such as graft or flap)
7. Other disease according to investigator's judgment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who present to the emergency department or Plastic Surgery clinic after a hand trauma causing a metacarpal or phalangeal fracture.
Sampling Method: Probability Sample
Enrollment: 1042 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Infection rate post closed reduction internal fixation | 12 weeks post fixation
  The rate of infections after K-wire fixation of hand fractures. K-wire infection will be diagnosed if two of the three following criteria are met: i) surrounding cellulitis greater than 5mm of diameter around K wire site (more than normal inflammation) ii) purulent drainage from the pin site and iii) bacteriologic evidence of infection (ie: positive cultures). X-ray evidence of osteomyelitis will also be considered for diagnosis of late infection.

SECONDARY OUTCOMES:
Complication rate post closed reduction internal fixation | 12 weeks post fixation
  The rate of other complications after K-wire fixation of hand fractures. These include issues such as malunion and nonunion.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Lalonde, MD, Principal Investigator — Horizon Health Network
Locations (15):
- Canada (14):
  - Univeristy of Calgary, Calgary, Alberta
  - Fraser Health, New Westminster, British Columbia
  - Lion's Gate Hospital, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Horizon Health Network, Saint John, New Brunswick
  - Memorial University, St. John's, Newfoundland and Labrador
  - St. Martha's Regional Hospital, Antigonish, Nova Scotia
  - Dalhousie University, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Univeristy of Ottawa, Ottawa, Ontario
  - University of Toronto, Toronto, Ontario
  - McGill University, Montreal, Quebec
  - University of Montreal, Montreal, Quebec
  - Saint-Hyacinthe, Saint-Hyacinthe, Quebec
- Philippine Orthopedic Center, Ma. Clara Corner Banawe Street, Quezon City, Philippines

IPD SHARING:
Plan to Share IPD: No
Patient information will be recorded using a corresponding number based on their order of presentation. The data will be presented or published as an average of all patients in the study.